CLINICAL TRIAL: NCT02880839
Title: Digital Navigation Enhances Cervical Pedicle Screw Placement Accuracy and Safety: A Randomized Controlled Trial
Brief Title: Digital Navigation Enhances Cervical Pedicle Screw Placement Accuracy and Safety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nantong University (Other)
Responsible Party: Principal Investigator, Junjie Guan, Attending Physician, Nantong University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NantongU_001
Record Dates: First submitted 2016-08-19; First posted 2016-08-26 (Estimated); Last update posted 2016-08-26 (Estimated); Status verified 2016-08

CONDITIONS: Cervical Spine Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Partial cervical lamina excision group (Experimental): Patients in the cervical lamina partial excision group underwent partial cervical lamina excision and cervical pedicle screw internal fixation.
  Interventions: Device: Partial cervical lamina excision group
- Pipeline-dredge discharge group (Experimental): Patients in the pipeline-dredge discharge group underwent pipeline-dredge discharge and cervical pedicle screw internal fixation.
  Interventions: Device: Pipeline-dredge discharge group
- Digital navigation group (Experimental): Patients in the digital navigation group underwent digital navigation-assisted cervical pedicle placement.
  Interventions: Device: Digital navigation group

INTERVENTIONS:
Device: Partial cervical lamina excision group — Patients with cervical fracture were assigned to undergo partial cervical lamina excision and cervical pedicle screw internal fixation.
  Arms: Partial cervical lamina excision group
Device: Pipeline-dredge discharge group — Patients with cervical fracture were assigned to undergo pipeline-dredge discharge and cervical pedicle screw internal fixation.
  Arms: Pipeline-dredge discharge group
Device: Digital navigation group — Patients with cervical fracture were assigned to undergo digital navigation assisted cervical pedicle screw placement.
  Other Names: Digital navigation system
  Arms: Digital navigation group

SUMMARY:
To compare the internal fixation results of three pedicle screw implantation methods and investigated the accuracy and safety of digital navigation-assisted pedicle screw placement.

DETAILED DESCRIPTION:
History and current status of related studies

The cervical pedicle is a tiny structure adjacent to important tissues including the spinal cord and vertebral artery. Cervical pedicle screw internal fixation is the conventional treatment for cervical spine fracture, and the technique provides acceptable internal fixation; however, current manipulation methods result in high pedicle screw penetration rates, a high risk of damage to peripheral vessels and nerves, and high rates of postoperative deformity. Improved techniques and minimally invasive methods such as transcutaneous pedicle screw implantation have been designed to effectively reduce surgery-related injury while maintaining the accuracy and safety of pedicle screw implantation. Unfortunately, there is no unified standard regarding implantation of cervical pedicle screws, and many pedicle screw implantation methods are used including partial cervical lamina excision and pipeline-dredge discharge. However, both of these techniques are clinically limited because of poor maneuverability. Digital navigation is an emerging technique based on the discrete-accumulation principle. The technique integrates computer methods, numerical control, laser and new materials, and provides a new digital technique for confirming the location and orientation of cervical pedicle screws, ensuring safe surgical operation.

Features different from other related studies

Previous studies focused primarily on investigating the curative effects of pedicle screw implantation in cervical spine fracture. To the best of the investigators knowledge, there are no studies of cervical spine fracture treatment by digital navigation-assisted cervical pedicle screw placement before June 2006 in Web of Science. The investigators located two similar articles (Cervical Spondylotic Myelopathy Surgical Trial (identifier: NCT02076113) and Slotted Hole Versus Fixed Hole C-Tek (identifier: NCT00585923)) in a search of ClinicalTrials.gov up to June 2006. The outcome measures in these two studies included bony fusion Short Form 36 and the physical component score. In contrast to these two studies regarding inclusion criteria and grouping, the investigators study was designed to investigate the accuracy and safety of digital navigation-assisted cervical pedicle screw placement, hoping to provide valuable quantitative evidence for the clinical application of this technique.

Adverse events

Possible adverse events included any expected or unexpected symptoms. If severe adverse events occurred, their details including the date of occurrence and measures taken to treat the adverse events were reported to the principal investigator and the institutional review board within 24 hours.

Data collection, management, analysis and open access

Data collection: Case report forms with demographic data, disease diagnosis, accompanying diseases, drug allergy history, and adverse events were collected, processed using Epidata software (Epidata Association, Odense, Denmark), collated, and then recorded electronically by data managers using a double-data entry strategy.

Data management: The locked electronic database was accessible and locked only by the project manager, and was not altered. Paper and electronic data regarding screening, informed consent, and clinical outcomes have been preserved at the Affiliated Hospital of Nantong University, China.

Data analysis: The electronic database was statistically analyzed by a professional statistician who created an outcome analysis report that was submitted to the lead researchers. An independent data monitoring committee supervised and managed the trial data, ensuring a scientific and stringent trial to yield accurate and complete data.

Data open access: Anonymized trial data was published at http://www.figshare.com.

Statistical analysis

Statistical analysis was performed by a statistician using SPSS 19.0 software (SPSS Inc.) and followed the intention-to-treat principle. Normally distributed measurement data was expressed as mean, standard deviation, and minimums and maximums. Non-normally distributed measurement data were expressed as lower quartile (q1), and median and upper quartile (q3). The Kruskal-Wallis H-test was used to compare the visual analogue scale spine scores among the three groups, and Fisher's exact test was used to compare the degree of bony fusion of the atlantoaxial joint and the incidence of adverse reactions. P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Fracture of the posterior column of the cervical spine or fracture of the anterior-posterior column of the cervical spine without severe vertebral body injury
* Non-traumatic cervical lamina destabilization, including metastatic tumor and rheumatoid arthritis
* Kyphotic deformity after cervical lamina resection
* Segmental destabilization after nerve root or spinal cord decompression
* Subjected to revision after anterior cervical spine surgery
* Scheduled to undergo internal fixation by cervical pedicle screw
* Age approximately 62 years
* Either sex
* Provision of signed informed consent to participate in the trial

Exclusion Criteria:

* Cervical pedicle injury resulting from trauma or tumor
* Severe osteoporosis
* Anatomical variation of the vertebral artery
* Unable or declined to proceed with internal fixation by pedicle screws

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
the penetration degree of the cervical pedicle screws | 12 months after internal fixation
  According to whether screws penetrated the pedicle and the degree of penetration, screw insertion was graded in three levels: grade I, pedicle screws do not penetrate the pedicular cortex; grade II, screw threads penetrate the cortex at the isthmic portion of the pedicle (no more than 1/4 length of the screw diameter); grade III, screws obviously penetrate the cortex at the isthmic portion of the pedicle (> 1/4 length of the screw diameter) with risk of peripheral nerve and vessel injury, and poor stabilization of the internal fixation.

SECONDARY OUTCOMES:
bony fusion rate of the atlantoaxial joint | 12 and 36 months after internal fixation
  To evaluate fracture healing. Bone fusion rate in the atlantoaxial joint was calculated as the percentage of patients with bony fusion of the atlantoaxial joint divided by the total patient number in each group.
Visual analogue scale spine score | prior to and 12 and 36 months after internal fixation
  To evaluate cervical neck pain. The visual analogue scale spine score ranges
American Spinal Injury Association Classification | prior to and 12 and 36 months after internal fixation
  To evaluate improvements in neurological function
incidence of adverse events | 12 and 36 months after internal fixation
  To evaluate the safety of each pedicle screw implantation method. The incidence of adverse events was calculated as the percentage of patients developing adverse events divided by the total patient number in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Junjie Guan, Master, Principal Investigator — Affiliated Hospital of Nantong University

IPD SHARING:
Plan to Share IPD: Undecided